CLINICAL TRIAL: NCT05505253
Title: Alfacalcidol Supplementation on Levator Ani Muscle Strength of Menopausal Pelvic Organ Prolapse Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OBGY-202206.03.
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: Alfacalcidol; MyoD expression; pelvic organ prolapse; vitamin D receptorr; levator ani muscle strength
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — alfacalcidol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alfacalcidol (Active Comparator): Alfacalcidol 0.5 mcg orally given for 3 months
  Interventions: Drug: Alfacalcidol 0.0005 MG
- Control (Placebo Comparator): Placebo given orally for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alfacalcidol 0.0005 MG — Alfacalcidol 0.5 mcg is given orally for 3 months, then vitamin D3 and vitamin D receptor levels are measured
  Arms: Alfacalcidol
Drug: Placebo — Placebo drug is given orally for 3 months, then vitamin D3 and vitamin D receptor levels are measured
  Arms: Control

SUMMARY:
This is a study performed to evaluate the role of vitamin D supplementation on the strength of levator ani muscle in menopausal women with pelvic organ prolapse

DETAILED DESCRIPTION:
Forty eight POP women were divided into experimental and control groups in this quasi-experimental study. The experimental group was given 0.5 mcg alfacalcidol orally for three months. We measured levator ani muscle strength, serum 25-hydroxy-vitamin D3 levels, and serum Vitamin D Receptor (VDR) levels at zero months and three months preoperative. Enzyme-linked immunosorbent assay (ELISA) assessed VDR and myoblast determination protein 1 (MyoD) protein expressions in levator ani muscle surgical biopsies.

ELIGIBILITY:
Inclusion Criteria:

* patients with pelvic organ prolapse stages III and IV who underwent surgery at menopausal age
* normal BMI
* initial serum vitamin D levels <30 ng/mL

Exclusion Criteria:

* comorbidities (chronic cough, conspitation)
* vitamin D metabolism or immune system interfering diseases or drugs specific routine medications such as anticonvulsants, statin, fibrate or orlistat
* history of vitamin D supplementation within the last month

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D3 levels | 3 months
  Vitamin D3 levels measured using lab tests
Vitamin D receptor levels | 3 months
  Vitamin D receptor levels as assessed by ELISA
Levator ani muscle strength | 3 months
  Levator ani muscle strength as measured using anometry

CONTACTS AND LOCATIONS:
Overall Officials: RM Sonny Sasotya, Ph.D., Principal Investigator — Universitas Padjadjaran
Locations (1):
- Universitas Padjadjaran, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient data are available upon written request to the authors
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: until 31 December 2026
Access Criteria: Access will be given upon written request to the authorrs

REFERENCES:
- [Result] Zhang L, Quan M, Cao ZB. Effect of vitamin D supplementation on upper and lower limb muscle strength and muscle power in athletes: A meta-analysis. PLoS One. 2019 Apr 30;14(4):e0215826. doi: 10.1371/journal.pone.0215826. eCollection 2019. PMID 31039170
- [Result] Latham CM, Brightwell CR, Keeble AR, Munson BD, Thomas NT, Zagzoog AM, Fry CS, Fry JL. Vitamin D Promotes Skeletal Muscle Regeneration and Mitochondrial Health. Front Physiol. 2021 Apr 14;12:660498. doi: 10.3389/fphys.2021.660498. eCollection 2021. PMID 33935807